CLINICAL TRIAL: NCT04697758
Title: Phase 1/2a Study of the Safety and Bioactivity of AXT-107 in Subjects With Diabetic Macular Edema (DME)
Brief Title: Safety and Bioactivity of AXT107 in Subjects With Diabetic Macular Edema
Acronym: CONGO
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Adverse Events
Sponsor: AsclepiX Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AXT107-CS101
Record Dates: First submitted 2020-12-17; First posted 2021-01-06 (Actual); Results first posted 2024-03-22 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Diabetic Macular Edema (DME)
Keywords: AsclepiX; macular edema; DME; eye diseases; retinal diseases; AXT107; diabetes; duration of action; dose escalation; diabetic retinopathy; retinal degeneration
MeSH Terms: conditions — Macular Edema; Eye Diseases; Retinal Diseases; Diabetes Mellitus; Diabetic Retinopathy; Retinal Degeneration | interventions — AXT107

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Low Dose (Experimental): AXT107 0.1 mg/eye
  Interventions: Drug: AXT107 0.1 mg
- Mid Dose (Experimental): AXT107 0.25 mg/eye
  Interventions: Drug: AXT107 0.25 mg
- High Dose (Experimental): AXT107 0.5 mg/eye
  Interventions: Drug: AXT107 0.5 mg

INTERVENTIONS:
Drug: AXT107 0.1 mg — Single intravitreal injection of AXT107 0.1 mg/eye
  Other Names: Gersizangatide
  Arms: Low Dose
Drug: AXT107 0.25 mg — Single intravitreal injection of AXT107 0.25 mg/eye
  Other Names: Gersizangatide
  Arms: Mid Dose
Drug: AXT107 0.5 mg — Single intravitreal injection of AXT107 0.5 mg/eye
  Other Names: Gersizangatide
  Arms: High Dose

SUMMARY:
This study is an open-label, dose-escalating, 48-week study assessing the safety, tolerability, bioactivity and duration of action of a single intravitreal injection of 0.1 mg, 0.25 mg, or 0.5 mg AXT107 in approximately 18 subjects (up to 6 subjects per dose) with Diabetic Macular Edema (DME).

DETAILED DESCRIPTION:
Upon providing informed consent, subjects will be sequentially enrolled into the study. Decision regarding dose escalation will be based on the recommendation from the Data Monitoring Committee (DMC). The first 3 eligible subjects will receive the low dose of AXT107 injection. After the 3 low dose subjects complete a 7-day follow-up, the DMC will review their safety data. If an acceptable safety profile is determined by the DMC, 3 additional subjects will be enrolled to receive the mid dose of AXT107 injection. Upon completion of a 7-day follow-up, review of the safety data, and determination of an acceptable safety profile by the DMC for the mid dose subjects, 3 additional subjects will be enrolled to receive the high dose of AXT107 injection.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age or older with diabetic macular edema (DME) diagnosis secondary to diabetes mellitus Type 1 or 2
* Best corrected visual acuity (BCVA) Early Treatment Diabetic Retinopathy Study (ETDRS) letter score of 65 to 23 in the study eye
* Willing and able to comply with clinic visits and study-related procedures
* Provide signed inform consent

Exclusion Criteria:

* Any signs of high risk proliferative diabetic retinopathy in the study
* Previously-treated patients who are not responders to anti-VEGF
* Panretinal laser photocoagulation within 6 months and macular laser photocoagulation with 3 months of screening in the study eye

Note: Other inclusion/exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2020-12-10 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amir Shojaei, PhD, Study Director — Asclepix Therapeutics
Locations (10):
- United States (10):
  - AsclepiX Investigative Site, Gilbert, Arizona
  - AsclepiX Investigative Site, Los Angeles, California
  - AsclepiX Investigative Site, St. Petersburg, Florida
  - AsclepiX Investigative Site, Boston, Massachusetts
  - AsclepiX Investigative Site, Reno, Nevada
  - AsclepiX Investigative Site, Eugene, Oregon
  - AsclepiX Investigative Site, Philadelphia, Pennsylvania
  - AsclepiX Investigative Site, Abilene, Texas
  - AsclepiX Investigative Site, McAllen, Texas
  - AsclepiX Investigative Site, The Woodlands, Texas

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: No participants were assigned to the "High Dose" Arm/Group" due to adverse events observed in the "Low Dose" and "Mid Dose" groups.
Period: Overall Study
Arm/Group | Low Dose | Mid Dose | High Dose
Started | 3 | 3 | 0
Completed | 3 | 3 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Enrollment was closed after mid dose cohort were enrolled. The study only enrolled 6 subjects.
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Dose | Mid Dose | Total
Number analyzed (Participants) | 3 | 3 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 0 | 3
  >=65 years | 0 | 3 | 3
Age, Continuous [Mean (Full Range); unit: years] | 58.3 [55 to 62] | 73.3 [71 to 75] | 65.8 [55 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 2 | 3 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 2 | 5
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Safety as Assessed by Incidence of Adverse Events (AEs)
Description: Incidence of ocular (study eye) and systemic AEs
Time Frame: Screening to Week 48
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose | Mid Dose
Number analyzed (Participants) | 3 | 3
Participants
  Serious Ocular Adverse Event Treatment Related | 2 | 1
  Serious Non-Ocular Adverse Event Not Related to treatment | 1 | 0

ADVERSE EVENTS:
Time Frame: 48 weeks
Arm/Group | Low Dose | Mid Dose
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 3/3 | 1/3
Other Adverse Events (participants affected / at risk) | 2/3 | 1/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Dose (N=3) | Mid Dose (N=3)
Ocular Hypertension (Eye disorders) | 1 (1) | 1 (1)
Glaucoma (Eye disorders) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) — Non-Ocular
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Dose (N=3) | Mid Dose (N=3)
Vitreous Floaters (Eye disorders) | 2 (3) | 1 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-31): https://cdn.clinicaltrials.gov/large-docs/58/NCT04697758/Prot_SAP_001.pdf